CLINICAL TRIAL: NCT07124026
Title: Postural Characteristics and Body Composition in Adolescents: A Generation Z Perspective - Alarming Rates of Thoracic Hyperkyphosis
Brief Title: Posture and Body Composition in Gen Z Adolescent
Status: Completed | Type: Observational
Sponsor: Ordu University (Other)
Collaborators: Balikesir University (Other); Cukurova University (Other); Gazi University (Other)
Responsible Party: Principal Investigator, FUAT YUKSEL, Dr., Ordu University
Other Study IDs: 2020-18
Record Dates: First submitted 2025-08-08; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Posture Disorders in Children
Keywords: Adolescent posture; Thoracic hyperkyphosis; Body composition

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Underweight Group: BMI-for-age < 5th percentile
  Interventions: Other: No Intervention: Observational Cohort
- Normal Weight Group: BMI-for-age between 5th-85th percentile
  Interventions: Other: No Intervention: Observational Cohort
- Overweight Group: BMI-for-age ≥ 85th percentile
  Interventions: Other: No Intervention: Observational Cohort

INTERVENTIONS:
Other: No Intervention: Observational Cohort — No intervention

SUMMARY:
This study aims to explore the relationship between posture and body composition in adolescents from Generation Z (born between 2002 and 2005). It was conducted as a cross-sectional study at a high school in Ankara, Turkey. A total of 572 students between the ages of 14 and 17 were included.

Researchers used photographic analysis to measure head, neck, and shoulder posture, as well as a digital inclinometer to assess the curvature of the upper spine (thoracic kyphosis). Body composition-such as body fat percentage, fat-free mass, and body mass index (BMI)-was evaluated using a bioelectrical impedance analyzer.

All participants and their parents provided informed consent. After data collection, participants attended an educational seminar about posture and healthy habits. The study was approved by the Gazi University Ethics Committee and conducted in accordance with the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents born between 2002-2005.
* No history of spinal surgery, neurological, or musculoskeletal disorders.

Exclusion Criteria:

* Presence of congenital/post-traumatic spinal deformities.
* Inability to stand independently for measurements.

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Adolescents
Sampling Method: Probability Sample
Enrollment: 572 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2020-02-15 (Actual); Study Completion 2021-11-15 (Actual)

PRIMARY OUTCOMES:
Thoracic kyphosis angle | Single assessment (day 1 of measurement)

SECONDARY OUTCOMES:
Craniovertebral angle | Single assessment (day 1 of measurement)
Sagittal shoulder angle | Single assessment (day 1 of measurement)
Body composition (BMI, fat%) | Single assessment (day 1 of measurement)

CONTACTS AND LOCATIONS:
Locations (1):
- Ordu University, Ordu, Altinordu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
**Data**: De-identified posture measurements, body composition data.
Time Frame: - **Timeframe**: Available after 6 months of publication.
Access Criteria: Contact PI with a valid research proposal. - **Restrictions**: Ethics committee approval require